CLINICAL TRIAL: NCT04169360
Title: Safety and Preliminary Efficacy of ANS-6637 to Reduce Drug Craving and Harm in People With Opioid Use Disorder
Acronym: SEARCH
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The FDA determined that there is not adequate safety information to continue clinical investigations using ANS-6637 and Amygdala Neurosciences, the product company of ANS-6637, is no longer pursuing research with this compound.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Sarah Kattakuzhy, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00088649
Record Dates: First submitted 2019-11-05; First posted 2019-11-19 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — ANS-6637

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ANS-6637 (Experimental): ANS-6637 600mg once daily for 12 weeks
  Interventions: Drug: ANS-6637
- Placebo arm (Placebo Comparator): Placebo 600 mg once daily for 12 weeks
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: ANS-6637 — White, oblong 300 mg tablet
  Arms: ANS-6637
Drug: Placebo oral tablet — White, oblong 300 mg tablet
  Arms: Placebo arm

SUMMARY:
This is a double blind, placebo controlled, randomized trial to evaluate the safety and preliminary efficacy of ANS-6637 in adults with opioid use disorder with and without opioid agonist therapy. Patients will be randomized to two arms: (1) ANS-6637 for three months vs (2) Placebo for three months. Subjects will subsequently be followed for an additional one month post treatment.

DETAILED DESCRIPTION:
This is a double blind, placebo controlled, randomized trial to evaluate the safety and preliminary efficacy of ANS-6637 in adults with opioid use disorder with and without opioid agonist therapy. At screening, after providing consent, participants will be evaluated to ensure criteria for opioid use disorder by DSM V criteria is met, and whether the subject is receiving opioid agonist therapy will be determined. Participants will undergo a medical evaluation (including medical history, laboratory tests and EKG evaluation) to establish baseline medical and psychiatric diagnosis in order to ensure safety of participation. Once enrollment criteria are met, patients will be randomized in a blinded fashion to ANS-6637 or placebo, stratified by site and form of opioid agonist therapy. On Day 0, patients will be initiated on ANS-6637 vs. placebo according to randomization group. Subjects will be seen twice per week for two weeks, followed by weekly for two weeks, and then monthly for two months.

ELIGIBILITY:
Inclusion Criteria:

* Must have the ability to understand and must personally sign a written informed consent form, which must be obtained prior to initiation of study procedures.
* Must be between 18 and 65 years of age, inclusive.
* Must have the diagnosis of opioid use disorder by DSM (Diagnostic and Statistical Manual of Mental Disorders) V criteria of at least mild severity
* Must have a total score of 9 or greater (out of a total of 30) on the Opioid Craving Scale at screening
* If on opioid agonist therapy, must be on Opioid Agonist Therapy (OAT) medication for a minimum of six months prior to screening.
* If on medication for depression or anxiety, must be on a stable dose for a minimum of two months prior to screening.
* Must be able to take oral medication and be willing to adhere to the medication regimen
* Must agree to utilize the "AI Cure" platform, either on their personal phone or on a supplied device, for both daily video adherence monitoring as well as daily questionnaires for the entire study duration.
* Male subjects must refrain from sperm donation throughout the study period, and continuing for at least 90 days following the last dose of study drug.
* Subjects must refrain from blood donation throughout the study period, and continuing for at least 30 days following the last dose of study drug.
* Must be willing to comply with contraception guidelines: The fetal risks associated with ANS-6637 are not known, but pre-clinical animal data demonstrate some risk. Subjects must agree not to become pregnant or impregnate a female. Females of childbearing potential must have a pregnancy test at screening and baseline (Day 0). If pregnancy occurs or is suspected to occur, study staff must be notified immediately. For the duration of the study, subjects or female partners of childbearing potential must use one of the following, unless she is surgically sterile, post-menopausal, or partner is surgically sterile: oral contraceptives (OCP), contraceptive sponge, patch double barrier (diaphragm + spermicide or condom + spermicide), intrauterine device (IUD), etonogestrel implant, injection, hormonal vaginal contraceptive ring or complete abstinence
* Must be willing and able to comply with all study requirements and plan to attend all clinic visits.

Exclusion Criteria:

A subject will be ineligible for this study if 1 or more of the following criteria are met:

* Clinically significant AND grade 2 or higher abnormal laboratory values at screening, as determined by principal investigator
* Aspartate transaminase (AST) or Alanine transaminase (ALT) > 2.5 x upper limit of normal or total bilirubin > 1.6 x the upper limit of normal
* Creatinine clearance < 60 mL/min/1.73m2 by Chronic kidney disease (CKD)-Epidemiology Collaboration (EPI) Score.
* Personal or family history of Parkinson's Disease
* Diagnosed major depression AND with current self-reported depression episode
* Diagnosed generalized anxiety disorder AND with current self-reported uncontrolled anxiety
* Current self-reported suicidal ideation
* Diagnosed liver disease, including untreated chronic Hepatitis C (defined as detectable Hepatitis C RNA), Hepatitis B (defined as positive HBsAg), and/or cirrhosis (defined as Fibrosis (FIB)-4 > 3.25 AND confirmed by Fibroscan or Fibrosure)
* Diagnosed Human Immunodeficiency Virus (HIV) AND detectable viral load > 40 copies/mL
* Diagnosed moderate or serious dementia Taking any of the following medications in the last 6 months: dopamine agonist, dopamine antagonist, anti-psychotic, anti-convulsant (except for benzodiazepines and gabapentin) or barbiturate
* Inability to obtain venous access for sample collection.
* Had a prior history of any severe adverse reactions to ethanol [e.g., flushing (noticeable redness of the neck or throat) and/or increased heart rate (subject reports sensation of increased heart rate or palpitations) after drinking alcohol].
* Known hypersensitivity to formulation excipients: microcrystalline cellulose, croscarmellose sodium, magnesium stearate, polyvinyl alcohol, titanium dioxide, polyethylene glycol, and talc.
* Have previously participated in an investigational trial involving administration of any investigational compound within 30 days prior to screening
* Have any unresolved legal issues that could jeopardize continuation or completion of the study, at the discretion of the principal investigator
* Have any serious or active medical, surgical, or psychiatric conditions which, in the opinion of the Investigator, would interfere with subject treatment, assessment, or compliance with the protocol.
* Are unable to comply with study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Number of Grade 3-4 events, Grade 2 Significant event | 16 weeks
  The number of Grade 3-4 adverse events, as defined by the Division of AIDS (DAIDS) Toxicity Table Version 2.1, July, 2017 as well as the number of Grade 2 events requiring medication interruption or deemed clinically significant by a study investigator

SECONDARY OUTCOMES:
Urine Drug Screen | 16 weeks
  Percentage opioid free period by urine drug screen
Opioid Craving | 16 weeks
  Opioid craving will be assessed using the Opioid Craving scale questionnaire. The questionnaire consists of three questions and each of these questions has a minimum value of 0 and a maximum value 10. A score of 0 on each question is the best outcome; a score of 10 on each question is the worst outcome.
Opioid Agonist Therapy (OAT) concentration | 16 weeks
  Serum concentration of buprenorphine or methadone
Self reported description of drug use (Self-reported frequency/quantity/mode of opioid use, self-reported use of other drugs, overdose and overdose death) | 16 weeks
  Self-reported frequency/quantity/mode of opioid use as well as self-reported use of other drugs will be gathered using the Drug Use Survey. Subjects will indicate frequency of opioid use by documenting the number of times they used an opioid during a given day. The quantity of opioids used will be determined by the dollar amount of opioids the subject reports they have consumed during that day. Subjects will also report mode of opioid use by indicating whether they are using opioids via injection, skin popping, snorting or oral. The Drug Use Survey will also ask subjects to report incidence of use of non-opioid substances. Incidence of overdose will be captured with the Naloxone questionnaire which asks, "since you last visit, have you experienced an overdose?". Incidence of overdose death will measured by the number of medical examiner confirmed deaths of study participants with cause of death listed as "overdose related to an opioid".

OTHER OUTCOMES:
Change in Darke HIV Risk Taking Behavior Survey Score | 16 weeks
  The Darke HIV Risk Taking Behavior Questionnaire will be administered to assess subject's self-reported risk taking behaviors. Total scores on the test range from 0 to 55, with higher scores indicating a greater degree of risk-taking behavior.
Change in HIV Test Result | 16 weeks
  An HIV test (fourth generation antigen/antibody test) will be administered and the results are reported as either positive or negative.
Change in Hepatitis C (HCV) RNA result | 16 weeks
  A Hepatitis C (HCV) RNA test will be administered. This test measures the quantity of detectable RNA which is measured in IU/ml.
Change in appetite | 16 weeks
  Self reported changes in appetite will be captured by the Adverse Event Survey. The survey will ask, "since your last visit, have you had an increase in your appetite or a decrease in your appetite?".

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Kattakuzhy, MD, Principal Investigator — Institute of Human Virology at the University of Maryland

IPD SHARING:
Plan to Share IPD: Yes
The investigator will share de-identified data with approved outside collaborators under appropriate agreements, at the time of publication or shortly thereafter.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available at the time of publication or shortly thereafter, and will be kept indefinitely.
Access Criteria: Will be determined by Principal Investigator